CLINICAL TRIAL: NCT00800553
Title: The Neural and Behavioral Correlates of How Donepezil Modulates Memory and Inhibitory Efficiency in the Context of 24 Hours of Sleep Deprivation
Brief Title: fMRI-behavioral Study of Cholinergic Augmentation With Donepezil in Healthy Sleep Deprived Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Michael WL Chee, MBBS, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CRT108999
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Sleep Deprivation
Keywords: sleep deprivation; fMRI; double blind crossover study
MeSH Terms: conditions — Sleep Deprivation | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- donepezil (Experimental): donepezil, 5 mg p.o. for approx 2 weeks
  Interventions: Drug: donepezil
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: donepezil — 5mg o.m. p.o. for approx. 2 weeks
  Other Names: Aricept
  Arms: donepezil
Drug: Placebo — 5mg of placebo for approx. 2 weeks
  Arms: placebo

SUMMARY:
The purpose of this study was to characterize how the anti-cholinesterase inhibitor (AChE-I) donepezil modulates brain regions involved in visual short-term memory, episodic memory and inhibitory efficiency following 24 hours of total sleep deprivation using fMRI as an additional marker for drug effect.

DETAILED DESCRIPTION:
Short-term total sleep deprivation (SD) can result in cognitive impairments (Durmer and Dinges, 2005) that contribute to industrial catastrophes, transportation accidents, and medical errors (Mitler et al., 1988; Dinges, 1995; Barger et al., 2006; Philip and Akerstedt, 2006). This has motivated the use of pharmacological countermeasures, the most widely used being caffeine (Bonnet et al., 2005). Functional imaging studies of sleep-deprived persons could provide information concerning the neural substrates associated with SD-induced cognitive decline and in addition, provide functional assays for assessing drug effects. However, despite the growing number of functional imaging studies involving SD (Chee and Chuah, 2008), neuropharmacological studies in this context are rare (Thomas and Kwong, 2006).

Impairment of attention in sleep-deprived persons (Lim and Dinges, 2008) is an important cognitive deficit that affects other 'higher' cognitive operations, for example, visual short-term memory (VSTM) (Chee and Chuah, 2007). VSTM is used in service of many higher cognitive operations and has a capacity limit (Luck and Vogel, 1997; Cowan, 2000) that has neuroimaging correlates (Linden et al., 2003; Majerus et al., 2007; Mitchell and Cusack, 2007). SD-induced decline in VSTM capacity has been shown to originate from depressed visual attention or visual processing (Chee and Chuah, 2007). This was inferred from observing state-dependent, but load-independent, attenuation of parieto-occipital activation elicited by two visual tasks in which memory and perceptual load were independently and parametrically varied. Critically, the load-independent manner in which SD affected parieto-occipital activation across the tasks signified that something more fundamental than memory was depressed.

We reasoned that the decline in attention/visual processing might arise from reduced noradrenergic and cholinergic drive, given that these neurotransmitters underlie the maintenance of wakefulness (Everitt and Robbins, 1997; Steriade and McCarley, 2005) as well as visuospatial attention (Everitt and Robbins, 1997; Phillips et al., 2000). Increasing cholinergic transmission may improve visual working memory by increasing the selectivity of perceptual processing in the visual cortex (Furey et al., 2000a). Other experiments on visual memory have suggested that behavioral benefit may be associated with increases in extrastriate (Furey et al., 2000a; Lawrence et al., 2002) and superior parietal (Mentis et al., 2001) regions. Conversely, cholinergic blockade using scopolamine may impair orienting responses that involve parietal regions (Davidson and Marrocco, 2000).

Of relevance to the present study, the concentration of cholinergic effects in the parieto-occipital region coincides with the locus of state effects in several functional imaging studies of short term memory (Habeck et al., 2004; Chee and Chuah, 2007; Lim et al., 2007) in sleep-deprived persons.

Collectively, these findings led us to hypothesize that SD-induced deficits in visual processing/attention might benefit from cholinergic augmentation. We anticipated that the neural correlates of such performance modulation could be tracked by observing task-related parieto-occipital activation. To evaluate these hypotheses, we conducted a double-blind, placebo-controlled, cross-over functional imaging study to characterize the effect of donepezil on healthy young adults. In this within-subjects design, volunteers were scanned four times, twice following a normal night's sleep and twice after 24 hours of total SD.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is able to read and understand the Subject Information Sheet and comply with protocol requirements, instructions and protocol-stated restrictions.
2. Prior to any screening procedures, the subject and the physician must have signed a study-specific Informed Consent Form. No study-related procedures may be performed before the physician has obtained written informed consent from the subject.
3. The subject is between 21 years to 35 years of age.
4. The subject has a BMI of between 18.5 kg/m2 to 32 kg/m2 and body weight ≥ 50 kg.
5. The subject is right-handed.
6. The subject has a resting pulse >40 bpm and <90 bpm (normal range). The subject has a resting systolic blood pressure of between 91 mmHg to 140 mmHg (supine normal range) and a resting diastolic blood pressure of between 51 mmHg to 90 mmHg (supine normal range).
7. The subject, in the opinion of the investigator, is in good health on the basis of a pre-study physical examination, medical history, vital signs, electrocardiogram (ECG), and the results of blood chemistry, haematology, and serology tests, and a urinalysis. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
8. The subject has habitual good sleeping habits: sleeping on average 6.5 to 9 hours each night in the past month.
9. Have regular sleeping hours whereby they sleep no later than 1 am and rise before 9 am each day.
10. Have no history of excessive daytime sleepiness or insomnia.
11. Score no greater than 22 on the Morningness-Eveningness scale [Horne and Ostberg, 1976].
12. If female, the subject must use a double barrier method of contraception (2 separate methods of contraception) from Screening until final discharge from the study. Oral contraceptives are not allowed.

Exclusion Criteria:

1. The subject has taken prohibited medication within 1 week (or 14 days if the drug is a potential enzyme inducer) or within 5 half-lives prior to first dosing for any medication ingested, whichever is longer) prior to first dosing, unless in the opinion of the investigator and sponsor, the medication will not interfere with the study procedures or compromise safety. Prohibited medication is any prescribed medication or over-the-counter (OTC) medication, including high-dose vitamins or dietary supplements, or any herbal medicine known to interfere with the metabolic CYP pathways, (e.g. St. John's Wort) or cognitive function (e.g. ginko). Paracetamol for mild analgesia will be permitted.
2. The subject has a significant history of drug or alcohol abuse, defined as an alcohol intake greater than 21 units per week or a history of drug abuse within the last 6 months, or a history of substance abuse deemed significant by the investigator. A unit of alcohol is defined as 250 mL of lager/beer, 100 mL of Wine, or 25 mL of spirits.
3. The subject has an orthostatic blood pressure reduction >20 mmHg (based on the difference of systolic blood pressure between supine and after standing for 1 minute).
4. The subject has been exposed to more than 3 new chemical entities (NCEs) within 12 months prior to the first dosing day, or participated in a trial with any drug within 84 days before the start of the study, or participated in a trial with a NCE within 112 days before the start of the study.
5. History or presence of hypersensitivity to the study drugs or drugs of this class (hyoscine, atropine, donepezil) or a history of other severe drug allergy or hypersensitivity which, in the opinion of the physician responsible, contraindicates their participation.
6. The subject has a serious illness, such as liver or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic, or metabolic disturbance or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
7. The subject has history or presence of peptic ulcer disease, cardiac arrhythmias, cardiac conduction abnormalities, asthma or obstructive pulmonary disease.
8. The subject has history or presence of psychiatric or neurological illness, obstructive sleep apnea, narcolepsy or periodic leg movements as ascertained by questionnaire.
9. If participation in the study will result in the subject having donated more than 1500 mL blood in the previous 12 months and where participation in study would result in donation of blood in excess of 500 mL within a 56 day period.
10. The subject smokes more than 10 cigarettes per day or uses other nicotine containing products equivalent to 10 cigarettes per day (for example, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) and is not able to refrain from using nicotine containing products during the complete study period.
11. The subject tested positive after screening or at baseline for drugs of abuse (opiates, methadone, cocaine, amphetamines, barbiturates, benzodiazepines, and cannabinoids).
12. Caffeine intake of greater than 5 drinks per day on average.
13. Presence of glaucoma or raised intraocular pressure based on medical history.
14. Has an abnormality on acoustic function.
15. The presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies.
16. The volunteer reports previous marked feelings of claustrophobia in enclosed environments.
17. Abnormal anatomical MRI as defined by a radiologist on pre-study screening e.g. tumours, evidence of stroke, localized white matter lesions, excessive atrophy (local or global), aneurysms, vascular malformations.
18. Subjects who cannot complete the neuropsychological test battery despite having undergone the training sessions.
19. The subject's QTc (using Bazett's correction) is equal or greater than 430 ms (at Screening) as read on the printout of the ECG produced by the ECG equipment and evaluated by the investigator.
20. The subject, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
fMRI signal change in response to cholinergic augmentation within the context of sleep deprivation | approx 1 month
behavioral changes (response accuracy in a visual short term memory task) | approx 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael WL Chee, MBBS, MRCP, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Cognitive Neuroscience Laboratory, Duke-NUS Graduate Medical School, Singapore, Singapore

REFERENCES:
- [Result] Chuah LY, Chee MW. Cholinergic augmentation modulates visual task performance in sleep-deprived young adults. J Neurosci. 2008 Oct 29;28(44):11369-77. doi: 10.1523/JNEUROSCI.4045-08.2008. PMID 18971479
- See also: Cognitive Neuroscience Lab Webpage — http://www.cogneuro-lab.org/